CLINICAL TRIAL: NCT01925079
Title: A Randomized and Controlled Study About the Impact of Intensive Education on Lipid Management in Patients With Acute Coronary Syndrome in China
Brief Title: Intensive Education on Lipid Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Junbo Ge (Other)
Collaborators: Fujian Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Xi'an Jiaotong University (Other); The Luhe Teaching Hospital of the Capital Medical University (Other)
Responsible Party: Sponsor-Investigator, Junbo Ge, Professor, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACS-lipid-2013
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; statins; LDL-C; intensive education
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Educational Group (Experimental): The Intensive Educational Group will receive 5 visits, including 2 visits via phone contacts. The expected dates for each visit will be stamped on the follow-up brochure for convenience. Patient education in this group includes routine education at discharge; 4 educational brochures, a calendar with health tips, and follow-up brochure with medical expert letter sent to patients at the day for discharge (baseline); and educational short messages through message platform once a week. Dosage and adjustment of statins, and concomitant medications in all the treated patients will be recorded.
  Interventions: Behavioral: Intensive Education
- Control Group (Sham Comparator): The Control Group will receive 3 visits and receive care as per usual practice by the treating doctor and a follow-up brochure without medical expert letter. Dosage and adjustment of statins, and concomitant medications in all the treated patients will be recorded. Blood lipid panel (4 items), hepato-renal functions, and creatine kinase will be examined; while, Morisky 8-item questionnaire will be used to evaluate medication compliance at outpatient visits. In addition, the occurrence of major cardiovascular events and AE/SAE will be collected during the study.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Intensive Education — Statin Treatment：The investigator will be suggested to increase the dose of atorvastatin according to guideline if a patient's LDL-C does not achieve target level.
  Patient education:
  1. Routine education at discharge.
  2. 4 education brochures will be delivered to patients.
  3. Calendar with healthy tips will be delivered to patients before discharge.
  4. A follow-up brochure with medical expert letter.
  5. A total of 24 specific short messages for ACS will be developed and sent to patients (one short message per week).
  6. Telephone follow ups will be performed according to a standard communication document.
  At discharge, patients will be given a brochure for future follow up.
  Arms: Intensive Educational Group
Other: Control — Statin Treatment：The recommended dosage of atorvastatin will be adjusted at the physician's discretion.
  Patient education:
  1. Routine education at discharge.
  2. A follow-up brochure without medical expert letter.
  At discharge, patients will be given a brochure for future follow up.
  Arms: Control Group

SUMMARY:
Among the patients with coronary heart disease, those with ACS (acute coronary syndrome) are extremely high-risk patients. Therefore, management outside hospital, especially the regular administration of drugs, is vital to prevent the recurrence of cardiovascular events. However, most patients often fail to stay on a long-term administration regimen, especially the administration of statins. According to the statistics, the average duration adhered with statin in patients with ACS is less than 3 months, use of statin at hospital discharge was only 80% and 65% in 6 month, with a very low LDL-C control rate (about 11% at 6 months), which poses a threat to the recurrence rate of cardiovascular events in patients with ACS.

It was found in previous studies that there were many factors influencing patients' compliance, in which patients' refusing to take medicine accounted for a higher proportion. It suggests that patient had not recognized the importance of long-term administration. Therefore, it is extremely important for physicians to strengthen patient education and regular follow-up visits during disease management. Moreover, the effectiveness of patient education during chronic disease management has already been proved in some studies abroad, and the interventional effect of multiple patient education process outweighs that of single approach education.

Thus, we intend to conduct a randomized and controlled study to explore the effect of multi-channel intensive patient education on LDL-C target achieving rate and statin adherence in patients with ACS in China.

ELIGIBILITY:
Inclusion Criteria:

1. The patients admitted to the hospital with a diagnosis of ACS including those for first consulting or with recurrence. The patient was prescribed atorvastatin (Lipitor®) by physicians in hospital;
2. The age of patient enrolled will be ≥18 years old;
3. The patient is able to understand and complete questionnaire.
4. The patients agree to accept follow-up visits, and willing to participate in patient education courses and sign informed consent form.

Exclusion Criteria:

1. The patient has contraindications to statins, such as active hepatic disease, patient has a history of intolerance or hypersensitivity to statins or has a history of prior rhabdomyolysis on a statin.
2. The patient who uses other statins except Lipitor® when discharged from the hospital;
3. Cardiac function class of the patient is class IV(NYHA);
4. The patient has a malignant tumor;
5. The patient has a severe arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2568 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-02 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
LDL-C target achieving rate | at Week 24 post-discharge

SECONDARY OUTCOMES:
LDL-C target achieving rate | at Week 12 post-discharge
the proportions of patients with statin persistence | at Week 12 post-discharge
the proportions of patients with statin persistence | at Week 24 post-discharge
statin compliance | at Week 12 post-discharge
statin compliance | at Week 24 post-discharge
the relationship of LDL-C target achieving rate and statin compliance | at Week 24 post-discharge
the discontinuation reason of statin therapy | at Week 24 post-discharge
the difference of LDL-C control rate and statin compliance | at Week 24 post-discharge
  To find the difference of LDL-C control rate and statin compliance between pre-specified sub-groups: PCI or non-PCI/male or female/age (≥65) or not/ having medical insurance or not/dyslipidemia history or not /MI (myocardial infarction) or UA (unstable angina)/different risk level according to TIMI/ patients for first consulting or patients with recurrence/ have received statin in the last 3 months or not.

OTHER OUTCOMES:
the major adverse cardiovascular events | at 24 weeks follow up

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Professor, Principal Investigator — Fudan University
Locations (5):
- China (5):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The 2nd affiliated hospital of harbin medical university, Harbin, Heilongjiang
  - Xi'an Jiaotong University College of Medicine, Xi’an, Shanxi
  - The Luhe Teaching Hospital of the Capital Medical University, Beijing
  - Shanghai Zhongshan Hospital, Shanghai